CLINICAL TRIAL: NCT01829906
Title: Evaluation of the Efficacy of Two Lifestyle Interventions for Suboptimal Weight Loss After Gastric Bypass Surgery
Brief Title: Suboptimal Weight Loss After Gastric Bypass Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: too few candidates for enrollment
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 321
Record Dates: First submitted 2013-04-09; First posted 2013-04-11 (Estimated); Last update posted 2017-10-04 (Actual); Status verified 2017-09

CONDITIONS: Obesity, Morbid
Keywords: weight loss; bariatric surgery; gastric bypass; health education; nutrition therapy; diet; exercise; cognitive therapy
MeSH Terms: conditions — Obesity, Morbid; Weight Loss; Health Education; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Outpatient group (Experimental): Multidisciplinary outpatient programme including both individual and group-based therapy. During the first visit, every patient will have an individual consultation with the dietician, physiotherapist and psychiatric nurse. After this, the patients will be followed up in groups every month for the first four months and every two months afterwards up to one year. The intervention will focus on nutritional education, healthy eating, increased physical activity levels (aiming initially at 10 minutes/day, then increasing to 30 minutes/day) and cognitive therapy.
  Interventions: Behavioral: Multidisciplinary outpatient programme
- Inpatient group (Experimental): Inpatient lifestyle programme offered at a rehabilitation center consisting of a "continuous care" weight loss program, with three intermittent stays (each with three-week duration) over a one year period.
  Interventions: Behavioral: Inpatient lifestyle programme

INTERVENTIONS:
Behavioral: Multidisciplinary outpatient programme
  Arms: Outpatient group
Behavioral: Inpatient lifestyle programme
  Arms: Inpatient group

SUMMARY:
Bariatric surgery is the only long-term established treatment for morbid obesity. However, some patients experience suboptimal weight loss after surgery and/or experience a significant weight regain. Unfortunately there are very few studies in this area and little is known about the causes for lack of success or the best approach to treat this group of patients. The main aim of this study is to compare the efficacy of two different lifestyle treatment programs in this group of patients: 1) Hospital-based outpatient program or 2) an inpatient treatment program consisting of 3 - 3-week stays at a rehabilitation center over a 1-year period. Secondary aim is to determine potential reasons for suboptimal weight loss after bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) >40kg/m2, or BMI>35kg/m2 with comorbidities
* healthy volunteers with suboptimal weight loss
* health with significant weight regain after Roux-n-Y Gastric Bypass, defined as failure to lose at least 40% Excess Weight Loss by 12 months postoperatively.

Significant weight regain: Regain of ≥15% of total weight lost after the first postoperative year.

Exclusion Criteria:

* Pregnancy
* enrollment in another obesity treatment
* previous revisional bariatric surgery
* planned bariatric surgery
* past or ongoing drug or alcohol abuse
* physical or mental impairment that interferes with the ability to comply to treatment
* history of severe psychological disorder
* history of severe eating disorder
* current medication known to affect appetite or induce weight loss

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Weight loss change | from baseline to 1 year
  Changes in body weight will be assessed at the end of the intervention (1 year)

SECONDARY OUTCOMES:
Risk factors | One year
  Risk factors: fasting plasma glucose and lipids (triglycerides, total cholesterol, HDL cholesterol) and blood pressure will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Bård Kulseng, md phd, Study Director — Norwegian University of Science and Technology
Locations (1):
- St. Olavs Hospital, Trondheim, Norway

REFERENCES:
- [Background] Amundsen T, Strommen M, Martins C. Suboptimal Weight Loss and Weight Regain after Gastric Bypass Surgery-Postoperative Status of Energy Intake, Eating Behavior, Physical Activity, and Psychometrics. Obes Surg. 2017 May;27(5):1316-1323. doi: 10.1007/s11695-016-2475-7. PMID 27914028